CLINICAL TRIAL: NCT05455073
Title: Evaluation of a Package of Nutrition Interventions to School-based Nutrition and Health Intervention for Adolescents in Bangladesh
Brief Title: Evaluation of School-based Nutrition Intervention for Adolescents in Bangladesh
Acronym: SNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition International (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); CDC Foundation (Other); Institute of Public Health and Nutrition, Ministry of Health and Family Welfare, Bangladesh (Unknown); Directorate of Secondary and Higher Education, Ministry of Education, Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NI-02-2019-SNAP
Record Dates: First submitted 2022-04-06; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-04

CONDITIONS: Anemia; Menstrual Hygiene Management; Improved Water, Sanitation and Hygiene (WASH)
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full package intervention arm (Experimental): * Dietary Supplement of Weekly Iron and Folic Acid (WIFA) Supplementation (containing 60 mg of elemental iron and 2800 µg of folic acid) and;
  * Associated behavior change intervention (BCI) to change the knowledge, attitudes, and practices of nutrition (including dietary diversity), IFA, deworming
  * Water, sanitation and hygiene (WASH) intervention: ensure availability (or provision) of water, sanitation, and hygiene supplies
  * Menstrual hygiene management (MHM) intervention: support for menstrual hygiene, including sale of menstrual products in schools
  * Associated behavior change intervention (BCI) to change the knowledge, attitudes, and practices (KAP) of WASH and menstrual hygiene management (MHM)
  Interventions: Dietary Supplement: Weekly Iron and Folic Acid Supplementation (WIFA); Combination Product: WASH; Combination Product: Menstrual Hygiene Management; Behavioral: Nutrition Behavior Change Intervention (BCI); Behavioral: MHM & WASH Behavior Change Intervention (BCI)
- Limited package intervention arm (Experimental): * Dietary Supplement of Weekly Iron and Folic Acid (WIFA) Supplementation (containing 60 mg of elemental iron and 2800 µg of folic acid; weekly school provision of WIFA tablets) and;
  * Associated behavior change intervention (BCI) to change the knowledge, attitudes, and practices of nutrition (including dietary diversity), IFA, deworming
  Interventions: Dietary Supplement: Weekly Iron and Folic Acid Supplementation (WIFA); Behavioral: Nutrition Behavior Change Intervention (BCI)
- Control (No Intervention): No intervention.

INTERVENTIONS:
Dietary Supplement: Weekly Iron and Folic Acid Supplementation (WIFA) — Weekly school provision of WIFA tablets to adolescent girls
  Other Names: Behavior Change Intervention
  Arms: Full package intervention arm; Limited package intervention arm
Combination Product: WASH — Ensure availability (or provision) of water, sanitation, and hygiene supplies for adolescent girls and boys
  Arms: Full package intervention arm
Combination Product: Menstrual Hygiene Management — Support for adolescent girls' menstrual hygiene
  Arms: Full package intervention arm
Behavioral: Nutrition Behavior Change Intervention (BCI) — Changing the knowledge, attitudes, and practices of nutrition (including dietary diversity), IFA, deworming
  Arms: Full package intervention arm; Limited package intervention arm
Behavioral: MHM & WASH Behavior Change Intervention (BCI) — Changing the knowledge, attitudes, and practices of WASH and menstrual hygiene management
  Arms: Full package intervention arm

SUMMARY:
Addressing the nutrition needs of adolescents could be an important initiative for breaking the vicious cycle of intergenerational malnutrition, chronic diseases and poverty. To respond to these diverse needs of adolescents, the Government of Bangladesh (GoB) in 2012, instituted a national policy for adolescent girls' weekly iron and folic acid (WIFA) supplementation in secondary schools to reduce anemia. Efforts are in place to roll out a national WIFA supplementation program for both in-school and out-of-school adolescent girls aged 10-19 years. Responding to the need to demonstrate the feasibility of such a new initiative before it is scaled-up, Nutrition International (NI) with funding support from the Government of Canada committed to providing technical and financial support to demonstrate to the GoB, the feasibility of a school-based delivery of nutrition interventions to improve the nutrition and health status of adolescents in Joypurhat and Sirajganj districts of Bangladesh. The project developed and began roll out of a multi-sectorial holistic and integrated nutrition approach consisting of both a nutrition-specific and nutrition-sensitive program model for improving the general health and nutrition of adolescents in schools. This was delivered in an integrated package for girls and boys including WIFA supplementation (girls only), promotion of improved water, sanitation and hygiene (WASH), behavior change interventions (BCI) on all topics, and support for menstrual hygiene management (MHM) for girls, including sale of menstrual products in schools. To evaluate the program, the GoB (Institute of Public Health and Nutrition, Ministry of Health and Family Welfare (IPHN) and The Directorate of Secondary and Higher Education, Ministry of Education (DSHE) and NI with technical assistance from the CDC Foundation and CDC planned process and outcome evaluations for the first year of the program's implementation.

DETAILED DESCRIPTION:
The outcome evaluation was a school (cluster)-based, randomized controlled trial with three equal size intervention arms, sampling adolescents, teachers, and student leaders in 75 selected schools. The study investigated the impact of the school-based program implemented in Joypurhat and aimed to examine the effectiveness and factors influencing scalability of using the secondary school platform to deliver WIFA co-packaged with WASH, MHM, and BCI to improve the nutrition and health status of adolescents in Bangladesh. The process evaluation sampled adolescents, teachers, and student leaders from 12 schools selected through convenience sampling for qualitative interviews, and determined whether the school-based program was implemented as intended, and why and how the intervention components worked to produce an impact - specifically, assessing the level of adherence.

ELIGIBILITY:
Inclusion Criteria:

* Randomly selected adolescent girl or boy
* Present on the day(s) of the survey
* Verbal assent and parental/guardian written consent
* School level headteacher, assigned teacher or student leader in the various grades

Exclusion Criteria:

* Girl or boy enrolled in grades other than grades 8 or 9
* Enrolled after random selection of participants

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3018 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration and anemia prevalence among adolescent girls | Up to 12 months
  Assessment of hemoglobin concentration and anemia prevalence among adolescent girls, using HemoCue® Hb-301 photometer
Iron and folate status, iron deficiency and folate insufficiency among adolescent girls | Up to 12 months
  a) Iron status and inflammation was assessed using a sandwich ELISA method, including 2 indicators of iron status (ferritin, sTfR) and 2 indicators of inflammation (C-reactive protein (CRP) and alpha 1-acid glycoprotein (AGP)); b) Folate status was assessed using a microbiological assay to test for red blood cell (RBC) folate and serum folate
Decrease morbidity among adolescents due to improved water, sanitation and hygiene (WASH) behaviour. | Up to 12 months
  Recall of morbidity symptoms over the past 3 days
Decrease barriers to menstrual hygiene management (MHM) for adolescent girls and thereby improve their school attendance | Up to 12 months
  In-school subsidized purchase of sanitary pads for menstruating girls

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition International, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demuyakor ME, Jalal C, Williams AM, Bouckaert KP, Whitehead RD Jr, Bhuiyan MM, Siraj S, Ara R, Pike V, Jefferds MED. Design, Methods, and Select Baseline Results from a School Nutrition Project for Adolescents in Bangladesh. Curr Dev Nutr. 2023 Mar 30;7(4):100070. doi: 10.1016/j.cdnut.2023.100070. eCollection 2023 Apr. PMID 37304846